CLINICAL TRIAL: NCT01227915
Title: RANDOMIZED CLINICAL EVALUATION OF EFFECTIVENESS COMPARISON BETWEEN DRUGS OPHTHALMOLOGICAL TOBRACORT® (TOBRAMYCIN + DEXAMETHASONE - LAB. UNIÃO QUÍMICA)AND TOBRADEX® (TOBRAMYCIN + DEXAMETHASONE - LAB. ALCON) IN REDUCING THE SIGNS AND SYMPTOMS OF ACUTE BACTERIAL CONJUNCTIVITIS
Brief Title: Effectiveness Comparison Between the Drugs TOBRACORT® and TOBRADEX® in Reducing the Signs and Symptoms of Acute Bacterial Conjunctivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clínica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TODUNI0610; Version 01
Record Dates: First submitted 2010-10-15; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Acute Bacterial Conjunctivitis
Keywords: SIGNS AND SYMPTOMS OF ACUTE BACTERIAL CONJUNCTIVITIS
MeSH Terms: interventions — Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Test (Experimental): tobramycin 0.3% + dexamethasone 1% - União Química Lab
  Interventions: Drug: Tobracort
- Comparator (Active Comparator): tobramycin 0.3% + dexamethasone 1% - Alcon Lab
  Interventions: Drug: Tobradex

INTERVENTIONS:
Drug: Tobracort — tobramycin 0.3% + dexamethasone 1%
  Arms: Test
Drug: Tobradex — tobramycin 0.3% + dexamethasone 1%
  Arms: Comparator

SUMMARY:
The primary objective of this study is to evaluate, through clinical parameters, the comparative efficacy between topical Tobracort ® (tobramycin 0.3% dexamethasone + 1% - Chemistry Lab Union) and TOBRADEX ® (tobramycin 0.3% dexamethasone + 1 % - Alcon Lab), using the percentage of improvement (sustained response rate) at the end of treatment.

DETAILED DESCRIPTION:
* Evaluation of signs and symptoms during treatment, with a record of individual scores for each parameter;
* Observation and statistical comparison of drug safety, by recording qualitative and quantitative parameters related to adverse effects occurring during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all study procedures and sign, by his own free will, IC;

  * Adult patients, regardless of gender, ethnicity or social status, with good mental health;
  * Patients who present at screening visit, a clinical picture of acute bacterial conjunctivitis diagnosed clinically.

Exclusion Criteria:

* Patients with clinical diagnosis of conjunctivitis due to any process other than bacterial infection, such as infections by fungi, protozoa, viruses, or allergic conjunctivitis;

  * Patients with a history or clinical diagnosis of other lesions that may affect the outcome, such as glaucoma, corneal ulcer or scars;
  * Patients with known hypersensitivity to any component of the study drug;
  * Concomitant use of ocular medication other than the study;
  * Patients who have made use of systemic anti-inflammatory hormone in the 30 days preceding inclusion;
  * Patients who have made use of systemic antibiotics in the 15 days preceding inclusion;
  * Pregnant or lactating women;
  * Being or having been treated for any type of conjunctivitis is less than 15 days, or have finished treatment at least 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness compared between drugs using the percentage of improvement (sustained response rate) at the end of treatment. | 7 days of treatment
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment.At the returns of 1 and 3 days, there will be a tolerance of +1 day, and the return of seven days, the tolerance will be ± 1 days. On each return, will be collected data on the efficacy and safety as defined in this protocol.

SECONDARY OUTCOMES:
Evaluation of signs and symptoms during treatment, with a record of individual scores for each parameter established. | 7 days of treatment.
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment.At the returns of 1 and 3 days, there will be a tolerance of +1 day, and the return of seven days, the tolerance will be ± 1 days. On each return, will be collected data on the efficacy and safety as defined in this protocol.
Statistical comparison of drug safety, by recording qualitative and quantitative parameters related to adverse effects occurring during treatment. | 7 days of treatment.
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment.At the returns of 1 and 3 days, there will be a tolerance of +1 day, and the return of seven days, the tolerance will be ± 1 days. On each return, will be collected data on the efficacy and safety as defined in this protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil